CLINICAL TRIAL: NCT03969173
Title: Determination of Best PEEP (Positive End-expiratory Pressure) in Anesthetized Infants in Terms of Prevention of Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2019-0224
Record Dates: First submitted 2019-05-15; First posted 2019-05-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pediatric Surgery
Keywords: Children undergoing pediatric general surgery or pediatric urology surgery

STUDY DESIGN:
Intervention Model Description: It is divided into the following three groups according to PEEP to be applied during anesthesia.
  Test group: PEEP6 group (6 cmH2O), PEEP9 group (9 cmH2O) control group: PEEP3 group (PEEP 3 cmH2O)
Masking Description: The physician who directly anesthetize the patient should not be aware of the patient's placement due to the nature of the study design and maintenance of anesthesia. The ultrasound examination of the patient's degree of atelectasis and data collection of cardiac index data was limited to a single anesthesiologist without knowing which group the patient is in. Blind cancellation is performed after data analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEEP3 (Active Comparator): The baseline atelectasis score is measured using sonography with no PEEP. And then, the baseline cardiac index is measured using transesophageal doppler for 5 minutes each with 3 cmH2O of PEEP. Apply PEEP (3 cmH2O) according to the patient's randomized group, and maintain the PEEP until the end of the operation.
  Interventions: Procedure: applying PEEP3
- PEEP6 (Active Comparator): The baseline atelectasis score is measured using sonography with no PEEP. And then, the baseline cardiac index is measured using transesophageal doppler for 5 minutes each with 3 cmH2O of PEEP. Apply PEEP (6 cmH2O) according to the patient's randomized group, and maintain the PEEP until the end of the operation.
  Interventions: Procedure: applying PEEP6
- PEEP9 (Active Comparator): The baseline atelectasis score is measured using sonography with no PEEP. And then, the baseline cardiac index is measured using transesophageal doppler for 5 minutes each with 3 cmH2O of PEEP. Apply PEEP (9 cmH2O) according to the patient's randomized group, and maintain the PEEP until the end of the operation.
  Interventions: Procedure: applying PEEP9

INTERVENTIONS:
Procedure: applying PEEP3 — The baseline atelectasis score is measured using sonography with no PEEP. And then, the baseline cardiac index is measured using transesophageal doppler for 5 minutes each with 3 cmH2O of PEEP.
  Apply PEEP (3 cmH2O) according to the patient's randomized group, and maintain the PEEP until the end of the operation.
  Arms: PEEP3
Procedure: applying PEEP6 — The baseline atelectasis score is measured using sonography with no PEEP. And then, the baseline cardiac index is measured using transesophageal doppler for 5 minutes each with 3 cmH2O of PEEP.
  Apply PEEP (6 cmH2O) according to the patient's randomized group, and maintain the PEEP until the end of the operation.
  Arms: PEEP6
Procedure: applying PEEP9 — The baseline atelectasis score is measured using sonography with no PEEP. And then, the baseline cardiac index is measured using transesophageal doppler for 5 minutes each with 3 cmH2O of PEEP.
  Apply PEEP (9 cmH2O) according to the patient's randomized group, and maintain the PEEP until the end of the operation.
  Arms: PEEP9

SUMMARY:
Purpose of research; to determine the appropriate positive end-expiratory pressure to minimize atelectasis during general anesthesia in infants.

Study design : Application of one pressure of PEEP among 3, 6, or 9 cmH2O during mechanical positive ventilation for general anesthesia to randomly assigned infants over 6 months to 13 months of age . Immediately after the start of anesthesia (PEEP=0) and before the end of anesthesia, the score of atelectasis is measured by lung ultrasonography with the standardized method. The scores at PEEP3, PEEP6, and PEEP9 will be compared to identify the appropriate PEEP at which atelectasis is the least likely to occur during anesthesia.

Medical Equipment : Ultrasonography with 6 - 13 MHz linear probe, Cardio-Q esophageal Doppler

The number of target subjects: According to the results of previous studies, the lung ultrasound score by ultrasonography at the end of anesthesia was 28.5 (IQR 21.8-37) without any recruitment (PEEP 0 cmH2O) (IQR 6-21.3). When PEEP of 5 cmH2O was maintained, the lung ultrasound score is 12.5 (IQR 6-21.3), which is lower than PEEP 0. It is assumed that the score at PEEP3 is 20, the score at optimal PEEP is 10, and the standard deviation is 11. Bonferroni correction is required for statistical analysis. In comparison between the two groups, alpha is used as the Bonferroni corrected alpha level of 0.05 / 3 = 0.017. The significance level alpha is fixed at 0.017 and the number of samples considering the 10% dropout rate when the power (1-β) is 80% is required to be 30 for each group.

Data analysis and statistical methods: Atelectasis score, cardiac index, peak inspiratory pressure, and dynamic compliance will be compared by t-test between groups(PEEP3 vs PEEP 6, PEEP 3 vs PEEP 9, PEEP 6 vs PEEP 9). P < 0.017 is going to be considered statistically significant.

DETAILED DESCRIPTION:
1. The selected pediatric patients undergo general anesthesia with the method commonly used in the operating room, and mechanical ventilation is applied to the patients after endotracheal intubation.
2. Within five minutes of the start of mechanical ventilation, the degree of baseline lung atelectasis is measured in anterior, lateral, and posterior regions of the upper and lower lungs of both lungs using transthoracic lung ultrasonography, ie, a total of 12 regions. Atelectasis is confirmed by the presence or absence of B-line and juxtapleural consolidation, grading to 0-3 according to severity. That is, the lung atelectasis score can be scored from 0 to 72 points.
3. After ultrasound examination, PEEP is applied in 3 cm H2O.
4. The cardiac index is measured using a transesophageal doppler for 5 minutes before (PEEP=3) and after each application of PEEP (3, 6, 9 cm H2O) according to a randomized, defined group of patients.
5. The applied PEEP is maintained until the end of the operation.
6. After the end of the operation, the score of the lung atelectasis is measured by the same method.
7. Patients who had atelectasis on ultrasonography are recruited three times for 3-5 seconds under 30 cmH2O pressure under the guideline of lung ultrasonography. The anesthesia is terminated by a conventional method and the patient is awakened. The patient is monitored at the recovery room and transferred to the general ward.

ELIGIBILITY:
Inclusion Criteria:

* 1. American Society of Anesthesiologists (ASA PS) I-II
* 2. pediatric general surgery or pediatric urology surgery under general anesthesia
* 3. over 6 months of age and less than 13 months of age
* 4. height and weight are 5-95% of peers

Exclusion Criteria:

* 1. Congenital heart or lung disease
* 2. hemodynamic unstable vital sign
* 3. bronchopulmonary dysplasia
* 4. laparoscopic surgery

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Lung atelectasis score after surgery | before the end of anesthesia
  Before the end of anesthesia, the degree of atelectasis is measured by lung ultrasonography and scored according to the standardized method. Comparison of the scores at PEEP3, PEEP6, and PEEP9 to identify the appropriate PEEP at which atelectasis is the least likely to occur during anesthesia.
  Lung atelectasis score:
  The 6-13 MHz linear probe of the ultrasonic device is applied perpendicular to the patient's ribs and evaluated using a 2 dimensional classic view. Transthoracic pulmonary ultrasound imaging is performed in 12 areas. One thoracic region is divided into 6 zones (caudal anterior, caudal lateral, caudal posterior, cranial anterior, cranial lateral, and cranial posterior) by three longitudinal lines (parasternal, anterior, and posterior axilla) and two axial lines (just above the diaphragm, nipple line). The degree of atelectasis(0-72 points) is the sum of the consolidation score (0-36 points) and the B-line score (0-36 points) in 12 areas.

SECONDARY OUTCOMES:
Cardiac index | During surgery, the cardiac index is measured using a transesophageal doppler for 5 minutes each before and after application of PEEP (3, 6, 9 cm H 2 O) according to the randomized, defined group of patients.
  The pediatric oesophageal doppler probe is used to compare the cardiac index for PEEP3 (baseline) and PEEP according to each group.
  Cardiac index:
  The CardioQ-ODM + can calculate Cardiac Index in Doppler flow mode. Cardiac Index relates the Cardiac Output to body surface area (BSA), thus relating heart performance to the size of the individual. The unit of measurement is litres per minute per square metre (l/min/m2).
  Cardiac Index = Cardiac Output/Body Surface Area The range of cardiac index is 2 to 6 L/min/m2.
Peak inspiratory pressure | During surgery, the cardiac index is measured using a transesophageal doppler for 5 minutes each before and after application of PEEP (3, 6, 9 cm H 2 O) according to the randomized, defined group of patients.
  Peak inspiratory pressure and dynamic compliance on the ventilator monitor during each PEEP are recorded.
Dynamic compliance | During surgery, the cardiac index is measured using a transesophageal doppler for 5 minutes each before and after application of PEEP (3, 6, 9 cm H 2 O) according to the randomized, defined group of patients.
  Peak inspiratory pressure and dynamic compliance on the ventilator monitor during each PEEP are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Lee JH, Kim HJ, Choi H, Lee JR. Optimal positive end-expiratory pressure to prevent anaesthesia-induced atelectasis in infants: A prospective, randomised, double-blind trial. Eur J Anaesthesiol. 2021 Oct 1;38(10):1019-1025. doi: 10.1097/EJA.0000000000001483. PMID 33720065